CLINICAL TRIAL: NCT07165509
Title: Neuro-Nutrition as Support for Physiological Function and Cognitive Abilities in Individuals With Down Syndrome, Autism Spectrum Disorder, and Attention-Deficit/Hyperactivity Disorder
Brief Title: Neuro-Nutrition to Support Physiological Function and Cognitive Skills in People With Down Syndrome, Autism Spectrum Disorder, and ADHD
Acronym: NEURODIET-DSAA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Elizabeth Guadalupe Ibarra Coronado (Network)
Collaborators: Universidad Nacional Autonoma de Mexico (Other)
Responsible Party: Sponsor-Investigator, Elizabeth Guadalupe Ibarra Coronado, Associate Research, Grupo de Neuroalimentación
Organization: Grupo de Neuroalimentación (Network)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CEI-000002-43; 157118 (Other: CONACYT (Mexico))
Record Dates: First submitted 2025-09-03; First posted 2025-09-10 (Actual); Last update posted 2025-09-10 (Actual); Status verified 2025-09

CONDITIONS: Down Syndrome; Autism Spectrum Disorder; Attention Deficit Hyperactivity Disorder (ADHD)
Keywords: Trisomy 21; ASD; ADHD; Neuro-nutrition; Structured diet; Dietary supplement; BRIEF; NEUROPSI Attention and Memory; Polysomnography; Sleep efficiency index; Apnea-hypopnea index; LDL cholesterol; C-reactive protein
MeSH Terms: conditions — Down Syndrome; Autism Spectrum Disorder; Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Intervention Model Description: Three-arm parallel study. Within each diagnostic cohort (Down syndrome, autism spectrum disorder, and ADHD), participants were assigned to one of three groups followed concurrently: (1) T-2 nutritional supplement (23 g twice daily) plus a structured dietary program; (2) structured diet only; or (3) no supplement and no structured diet (control). Age range 2-35 years; no crossover.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- T-2 Supplement + Structured Diet (Experimental): Participants receive the T-2 nutritional supplement (23 g twice daily) plus a structured dietary program. Arms run in parallel within each diagnostic cohort (Down syndrome, ASD, ADHD).
  Interventions: Dietary Supplement: T-2 Nutritional Supplement; Behavioral: Structured Dietary Program
- Structured Diet Only (Active Comparator): Participants follow the structured dietary intervention without the T-2 supplement.
  Interventions: Behavioral: Structured Dietary Program
- Control (No Intervention): Participants receive no T-2 supplement and no structured dietary program (usual diet).

INTERVENTIONS:
Dietary Supplement: T-2 Nutritional Supplement — Nutritional supplement labeled "T-2"; dose 23 g twice daily, as specified in the protocol. Used only in the arm "T-2 Supplement + Structured Diet."
  Other Names: Complemento Alimenticio T-2; T-2
  Arms: T-2 Supplement + Structured Diet
Behavioral: Structured Dietary Program — Rigorous, structured dietary intervention applied according to the study protocol. Used in the arms "T-2 Supplement + Structured Diet" and "Structured Diet Only."
  Other Names: Structured Diet; Neuro-Nutrition Diet Program
  Arms: Structured Diet Only; T-2 Supplement + Structured Diet

SUMMARY:
This study aimed to evaluate the impact of a specialized nutritional intervention on physiological performance, sleep quality, and cognitive abilities in individuals with neurodevelopmental disorders, specifically Down syndrome, autism spectrum disorders (ASD), and attention deficit disorder (ADD/ADHD). The intervention consisted of a modified diet protocol combined with an investigational nutritional formulation administered over a fixed intervention period. Outcomes included cognitive performance measures, sleep parameters, and selected physiological biomarkers.

DETAILED DESCRIPTION:
The Neuroalimentación protocol integrates dietary modification and targeted nutritional supplementation to support metabolic, cognitive, and physiological functions in populations with neurodevelopmental conditions. This interventional study was conducted as a longitudinal, prospective trial including participants diagnosed with Down syndrome, autism spectrum disorders, or ADHD. Participants received the intervention for a defined period, during which outcomes related to cognitive performance, physiological markers, and sleep quality were evaluated using standardized neuropsychological tests, polysomnography, and laboratory analyses.

The trial sought to determine whether such dietary and supplementation strategies could enhance functional performance and quality of life in these populations.

ELIGIBILITY:
Inclusion Criteria:

* Age 2-35 years at enrollment.
* Clinical diagnosis of Down syndrome (DS), Autism Spectrum Disorder (ASD/TEA), or Attention-Deficit/Hyperactivity Disorder (ADHD/TDAH). For DS, written karyotype confirmation; for ASD/ADHD, clinical criteria (DSM) and standardized scales per protocol (e.g., Conners).
* Parent/guardian able to provide written informed consent prior to study procedures.
* Willingness to comply with the assigned structured diet and/or supplement regimen and study visits.

Exclusion Criteria:

* Individuals outside 2-35 years or without DS/ASD/ADHD diagnosis.
* Healthy volunteers (no target neurodevelopmental condition).
* Inability or unwillingness to adhere to the dietary program and/or supplement (the team may request withdrawal for non-adherence as per protocol).
* Lack of informed consent from parent/guardian.

Ages: 2 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2022-03-26 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-05-01 (Actual)

PRIMARY OUTCOMES:
Change in Executive Function (BRIEF Global Executive Composite [GEC] T-score) | Baseline to 12 months
  Parent/caregiver-rated BRIEF; Global Executive Composite (GEC) T-score (normative mean 50, SD 10). Change is calculated as follow-up minus baseline; unit: T-score.

SECONDARY OUTCOMES:
Change in NEUROPSI Attention and Memory Total Standardized Score | Baseline to 12 months
  NEUROPSI Attention and Memory battery; standardized total score covering verbal/visual short- and long-term memory, episodic memory, attention/concentration, and motor skills; unit: standardized score/percentile per test manual.

OTHER OUTCOMES:
Sleep Efficiency Index (%) by Overnight Polysomnography | Baseline to 12 months
  Overnight polysomnography (≥8 h) recording EEG, EOG, EMG, airflow, respiratory effort, oximetry, etc. Sleep Efficiency Index defined as total sleep time divided by time in bed/recording × 100; unit: percent.
Apnea-Hypopnea Index (events/hour) by Polysomnography | Baseline to 12 months
  Number of respiratory alterations during sleep divided by total sleep time; unit: events/hour.
LDL Cholesterol (mg/dL) | Baseline to 12 months
  Fasting serum low-density lipoprotein cholesterol from standard blood chemistry panel; unit: mg/dL.
C-Reactive Protein (mg/L) | Baseline to 12 months
  Serum C-reactive protein as a marker of systemic inflammation; unit: mg/L.
Conners Parent Rating Scale-Revised: Hyperactivity Index T-score | Baseline to 12 months
  80-item parent-rated scale; Hyperactivity Index T-score per test manual; unit: T-score.

CONTACTS AND LOCATIONS:
Locations (1):
- Instituto Mexicano de Medicina Integral de Sueño, Mexico City, Mexico

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared because the informed consent approved by the research ethics committee did not authorize secondary sharing or posting of participant-level data. The dataset includes minors and sensitive health information; sharing would require re-consent and/or new ethics approval, which is not feasible for this completed study.

REFERENCES:
- [Background] Gioia GA, Isquith PK, Retzlaff PD, Espy KA. Confirmatory factor analysis of the Behavior Rating Inventory of Executive Function (BRIEF) in a clinical sample. Child Neuropsychol. 2002 Dec;8(4):249-57. doi: 10.1076/chin.8.4.249.13513. PMID 12759822
- [Background] MAHONEY FI, BARTHEL DW. FUNCTIONAL EVALUATION: THE BARTHEL INDEX. Md State Med J. 1965 Feb;14:61-5. No abstract available. PMID 14258950
- [Background] First MB, Pincus HA. The DSM-IV Text Revision: rationale and potential impact on clinical practice. Psychiatr Serv. 2002 Mar;53(3):288-92. doi: 10.1176/appi.ps.53.3.288. PMID 11875221
- [Background] Ostrosky-Solis F, Ardila A, Rosselli M. NEUROPSI: a brief neuropsychological test battery in Spanish with norms by age and educational level. J Int Neuropsychol Soc. 1999 Jul;5(5):413-33. doi: 10.1017/s1355617799555045. PMID 10439587
- [Background] Allik H, Larsson JO, Smedje H. Sleep patterns of school-age children with Asperger syndrome or high-functioning autism. J Autism Dev Disord. 2006 Jul;36(5):585-95. doi: 10.1007/s10803-006-0099-9. PMID 16617404
- [Background] Hering E, Epstein R, Elroy S, Iancu DR, Zelnik N. Sleep patterns in autistic children. J Autism Dev Disord. 1999 Apr;29(2):143-7. doi: 10.1023/a:1023092627223. PMID 10382134
- [Background] Accardo JA, Marcus CL, Leonard MB, Shults J, Meltzer LJ, Elia J. Associations between psychiatric comorbidities and sleep disturbances in children with attention-deficit/hyperactivity disorder. J Dev Behav Pediatr. 2012 Feb;33(2):97-105. doi: 10.1097/DBP.0b013e31823f6853. PMID 22261833
- [Background] Cotton S, Richdale A. Brief report: parental descriptions of sleep problems in children with autism, Down syndrome, and Prader-Willi syndrome. Res Dev Disabil. 2006 Mar-Apr;27(2):151-61. doi: 10.1016/j.ridd.2004.12.003. Epub 2005 Jun 21. PMID 15975763
- [Background] Bittles AH, Glasson EJ. Clinical, social, and ethical implications of changing life expectancy in Down syndrome. Dev Med Child Neurol. 2004 Apr;46(4):282-6. doi: 10.1017/s0012162204000441. No abstract available. PMID 15077706
- [Background] Billstedt E, Gillberg IC, Gillberg C. Autism after adolescence: population-based 13- to 22-year follow-up study of 120 individuals with autism diagnosed in childhood. J Autism Dev Disord. 2005 Jun;35(3):351-60. doi: 10.1007/s10803-005-3302-5. PMID 16119476
- [Background] Bieberich AA, Morgan SB. Brief report: affective expression in children with autism or Down syndrome. J Autism Dev Disord. 1998 Aug;28(4):333-8. doi: 10.1023/a:1026016804357. No abstract available. PMID 9711490

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2021-12-01): https://cdn.clinicaltrials.gov/large-docs/09/NCT07165509/Prot_ICF_000.pdf